CLINICAL TRIAL: NCT03485066
Title: Multimodal Associations of Human Brain Plasticity Investigated With Simultaneous PET/MR Imaging
Brief Title: Simultaneous PET/MR Imaging of Human Brain Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rupert Lanzenberger (Other)
Responsible Party: Sponsor-Investigator, Rupert Lanzenberger, Assoc.Prof. PD MD, Head of Neuroimaging Labs, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PSY-NIL-0005
Record Dates: First submitted 2017-04-28; First posted 2018-04-02 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Neuronal Plasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): 20 healthy participants, 4 week training of a challenging cognitive task (Tetris) between PET/MR measurements
  Interventions: Behavioral: Tetris
- Control (No Intervention): 20 healthy participants, no training between PET/MR measurements

INTERVENTIONS:
Behavioral: Tetris — The video game Tetris is a cognitively challenging task, which requires mental rotation, problem solving and fast visuo-spatial and motor coordination.
  Arms: Training

SUMMARY:
Background: Neuronal plasticity is the brain's ability to continuously adapt to experiences and learning of new skills. Although this affects multiple characteristics of the brain such as structure, function and metabolism, direct interactions between these aspects are largely missing.

Aim: Using recent advancements in neuroimaging we aim to identify novel relationships how neuronal plasticity is related across these characteristics.

Design: 40 healthy subjects will undergo two simultaneous PET/MR measurements at baseline and after 4 weeks. During the measurements a cognitively challenging task will be performed and the training group (20 subjects) will practice during the 4-week period.

Implications: We combine simultaneous PET/MR and novel task-specific PET imaging to study brain metabolism, structure and function in a single measurement session. This provides optimal sensitivity for assessment of multimodal neuroplasticity associations. Knowledge how cognitive training affects multiple characteristics of the brain will also increase our understanding of disorders like depression, dementia and brain injuries, since these are diagnosed with cognitive evaluations. Considering the vast usage of the applied imaging procedures in diagnosis and therapy monitoring, the thorough investigation of multimodal associations offers benefit for the interpretability of neuroimaging in clinical routine.

DETAILED DESCRIPTION:
Methodological details: Each subject will undergo two PET/MR examinations. Imaging will include PET as well as acquisition of structural and functional MRI. Task-specific glucose metabolism will be quantified with the radioligand [18F]FDG. Gray matter volume and white matter microstructure will be assessed with T1-weighted and diffusion weighted MRI, respectively. Functional imaging will focus on functional connectivity during rest and task as well as cerebral blood flow as acquired with ASL.

ELIGIBILITY:
Inclusion Criteria:

* Age range 21-30 years
* Right-handedness
* Willingness and competence to sign the informed consent form

Exclusion Criteria:

* History of or current physical, neurological or psychiatric disorder
* History of or current substance abuse or medication including antipsychotic, antidepressant and antianxiety agents
* Pregnancy or current breastfeeding
* Contraindications for MRI-scanning (e.g., metal implants, steel grafts, etc), including dental implants causing signal artifacts
* For subjects participating in earlier studies using ionizing radiation, the total radiation exposure of 30mSv over the last 10 years must not be exceeded, as specified in the Austrian legislation on radiation protection
* Regular players of the video game Tetris (3 years before scanning).
* Failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Training induced changes in imaging parameters | 4 weeks
  Imaging parameters are glucose metabolism ([18F]FDG PET), cerebral blood flow (arterial spin labeling MRI), functional connectivity (resting-state and task fMRI), gray matter volume (T1-weighted MRI) and white matter structure (diffusion weighted MRI)

SECONDARY OUTCOMES:
Cognitive performance | 4 weeks
  Training induced changes in performance of the video game (score per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, Assoc Prof, Study Director — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hahn A, Breakspear M, Rischka L, Wadsak W, Godbersen GM, Pichler V, Michenthaler P, Vanicek T, Hacker M, Kasper S, Lanzenberger R, Cocchi L. Reconfiguration of functional brain networks and metabolic cost converge during task performance. Elife. 2020 Apr 21;9:e52443. doi: 10.7554/eLife.52443. PMID 32314956
- See also: Neuroimaging Labs, Dept. of Psychiatry and Psychotherapy, Medical University of Vienna, Austria — http://www.meduniwien.ac.at/neuroimaging/